CLINICAL TRIAL: NCT06895694
Title: Investigation of the Effect of Education to Create Positive Hospital Perception in 8-10 Years Old Healthy Children
Brief Title: Creating a Positive Hospital Perception in Healthy Children Aged 8-10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Behice Ekici, Associate Professor, PhD, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/02-04
Record Dates: First submitted 2025-03-05; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Education
Keywords: Perception; Child; Hospital; Hospital Perception; Education

STUDY DESIGN:
Intervention Model Description: research and control group
Masking Description: research and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- research group (Experimental): After the first application of the scale, the children in the research group will be given "I am learning what kind of a place the hospital is" training using the direct expression method supported by a powerpoint presentation in line with the "Training content plan".
  Interventions: Other: examine the impact of education
- control group (No Intervention): Children in the control group were not trained.

INTERVENTIONS:
Other: examine the impact of education — Children in the research group were trained to create a positive hospital perception.
  Arms: research group

SUMMARY:
In this study, the effect of education in creating positive hospital perception for healthy children aged 8-10 years will be examined with a randomized controlled repeated measures design. All children between the ages of 8-10 attending Battalgazi Primary School in Sultanbeyli district of Istanbul province who meet the inclusion criteria (159 children in total) will be included. According to the results of the draw, 71 children will be included in the research group and 88 children will be included in the control group. The children assigned to the research group will be given the training prepared after the first measurement of the Hospital Perception Scale for Healthy Children. For the children in the control group, a second measurement will be made after the first application of the scale without any training. Children in the research and control groups will then be trained together. The content of the training will include introductions, what the hospital is like, what equipment and devices are in the hospital, who works in the hospital and what their duties are, what are the procedures performed in the hospital, how being in the hospital affects the child's life (sleep, play, eating and drinking, family, school, friends). The second measurement of the scale will be applied to the children in the research group after the training. The "Child Identifying Information Form" and "Informed Consent Form", which will be prepared by the researcher and the consultant for the children in the research and control groups to determine the age, gender, educational status, and previous hospital experiences of the child and his/her family, will be sent to the children and their parents one day before the training day and they will be asked to fill it out at home if they consent to participate in the study.

DETAILED DESCRIPTION:
Children are in the hospital for diagnosis, treatment, visits, short or long-term stays. Meanwhile, children; experiences unpleasant negative experiences such as pain, fear, anxiety, separation, restlessness, anger, regression, loneliness, frustration, introversion, and submission. During this period, a child who is admitted to hospital or admitted to hospital may feel a loss of control over his or her own health if he or she is examined, given blood or given medication without his or her will or consent. is stated in the literature that children under the age of 7 are afraid of unfamiliar people, new situations, abandonment and disability because their physiological, cognitive, emotional and social development has not reached a sufficient level. They also perceive hospitalization and hospital procedures as punishment for their bad behavior. Due to these developmental characteristics, these children; They may think that he will lose his best friend, stay away from his family, school and classes, and fail in his classes while he is hospitalized. During this period, the child who is admitted to the hospital or admitted to the hospital may think that he will lose control over his own body if he is examined, blood is taken, or medication is given against his will or consent. Some children may also think that they will have surgery, lose organs, become disabled, or even die. In addition, children who felt powerless and helpless in their past hospital experiences experienced more anxiety in their subsequent hospital experiences. They think that the child who experienced pain, aches, and fear in the past hospital experience will experience similar situations in the next experience It is stated that the child who has had a negative hospital experience in the past thinks that he will experience similar situations in his next experience. Research has shown that children aged 7-11 years perceive not being able to go to school or be with friends during their hospitalization as a negative experience and have high pain and procedural anxiety during phlebotomy. It was determined that children between the ages of 7-18 are afraid of injections (64.7%), being in a hospital environment (32.3%), staying away from home (3%), being injured (49.2%), having a bad disease (29.5%), death (13.1%), and taking medication (8.2%). In another study, it was determined that 70% of children under the age of 18 were afraid of vaccine injection. Studies have shown that negative childhood experiences will have negative physical and psychological health consequences; intense anxiety in the subsequent similar experience of children with hospital experience; they experience anxiety, fear and stress was determined. It was found that anxiety scores of children who were hospitalized for the first time were higher than those who were hospitalized more than once; anxiety scores increased with repeated hospitalizations and preoperative anxiety levels were high.

However, in the literature review, no study was found examining the hospital perception of sick or healthy children. In this study, the effect of education on positive hospital perception in healthy children aged 8-10 years will be examined. For this purpose, healthy children between the ages of 8 and 10 in the research group will be informed with the lecture method in line with the education program prepared according to their developmental levels and needs. After the briefing, it will be aimed to change these children's incorrect or incomplete information about the hospital and their negative perceptions of the hospital. Thus, in their subsequent experiences, children will adapt better to the diagnosis, treatment and care process, develop positive emotions and their recovery process will be shorter.

Methods:

This study will examine the effect of education to create positive hospital perception in healthy children aged 8-10 years with a randomized controlled repeated measures design.

The district and school where the research will be conducted will be randomly selected by lottery method after obtaining research permission from the ethics committee and Istanbul Provincial Directorate of National Education. The population of the research consisted of 215 children between the ages of 8-10 who attended the public Battalgazi Primary School in the Sultanbeyli district of Istanbul between Marth and May 2024.The sample size of the study was calculated with the G*Power 3.1.9.4 package program. Accordingly, for the two-tailed hypothesis to maximize the number of samples; margin of error α: 0.05, effect size (∆: 0.63) and power: 0.95; The minimum number of samples to be included in the study was calculated as 68 (total = 136) for each group. All children who met the inclusion criteria (159 children in total) were included in the sample to better reflect the population, to increase the generalizability of the research results, and to consider possible data loss. After collecting the research data, the power of the study was found to be 89% for 159 children, when alpha error was taken as 0.5%.

Procedures:

A simple randomization system was used for selection in the study. Children were assigned to the groups according to their class sections at school. For this purpose, firstly, the classes (2nd, 3rd and 4th grades) in which children aged 8-10 years without chronic health problems (A, C, D, E classes) were enrolled were determined together with the classroom teachers. Since the Hospital Perception Scale for Healthy Children (HPSHS) was used in healthy children, the class sections (2- B, 3-B, 4-B) in which children with chronic health problems (inclusion students) were enrolled were excluded from randomization.

The class sections (2-A, 3-A, 4-A, 2-C, 3-C, 4-C, 2-D, 3-D, 4-D, 2-E, 3-E, 4-E) were selected by lottery to be included in which group (research and control). The children in the first 3 classrooms (2-C, 3-D, 4-D) were assigned to the research group and the children in the second 3 classrooms (2-A, 3-A, 4-E) were assigned to the control group. All children in these classrooms who met the inclusion criteria (total = 159) were assigned to their groups. According to the results of the lottery, 71 children were included in the research group and 88 children were included in the control group.

Instruments:

In this study, data were collected with the Children's Introductory Information Form (CIIF) and the Hospital Perception Scale for Healthy Children (HPSHS). Children's Introductory Information Form (CIIF) and "I am Learning What a Hospital is Like" Training Content Plan were prepared by the researcher and consultant by scanning the relevant literature. All figures used in the training content were prepared by the researcher. Training content titles; Introduction, what is the hospital like, what equipment and devices are in the hospital, who works in the hospital and what are their duties, what are the procedures performed in the hospital, how does being in the hospital affect the child's life (sleeping, playing, eating and drinking, family, school, circle of friends).

Suitability of the educational content to the development level of children aged 8-10 and the research topic; It was evaluated by a child and adolescent psychiatrist (n = 1), a child development specialist (n = 1) and an academic pediatric nurse (n = 1). It was edited and finalized in line with the opinions and suggestions of experts.

Hospital Perception Scale for Healthy Children (HPSHS): This scale was developed by Ekici in 2023 to measure the hospital perception of healthy children in the 8-10 age group. The original language of the scale is Turkish and there are 25 scale items. At the beginning of the scale, there is an explanation of how to answer the scale items. Options for each item were created in a 3-point Likert type, depending on the child's level of participation in the item statement. Scoring of options; "I never think" is 0 points, "I sometimes think" is 1 point, and "I always think" is 2 points. There are no reverse scored items in the scale. The scale has a score range and cut-off points. The total score range of the 25-item scale varies between 0 and 50 points. The minimum score from the scale is "0" and the maximum score is "50". Interpretation of the total score of the scale; It is interpreted as "score between 0 and 24 = less negative hospital perception" and "score between 25 and 50 = more negative hospital perception". An increase in the scale score indicates that the child's negative perception of the hospital increases.

Through their classroom teachers, each child was given an "Informed Consent Form", "Child Introductory Information Form", and the HPSHS to be forwarded to their parents. In addition, the children's classroom teachers sent a brief information message to the parents of the children who were randomized. In this message; Examining the submitted forms and scale, if they approve the study (in writing); They were asked to fill out the "Child Introductory Information Form" together with the child, sign their consent, and send it back with their child the next day. In addition, it was stated that the HPSHS would be answered by the children before (the first measurement) and after (the second measurement) the "I am learning what kind of place a hospital is like" training at school. The first measurement of the "Hospital Perception Scale for Healthy Children" was carried out in the classrooms of the children in the research and control groups on a date deemed appropriate by the classroom teachers (March 26, 2024). Before the first measurement, the researcher first introduced himself when he went to the classrooms. Then, scale forms were distributed to each child, and they were asked to carefully read the 25 questions on the form and mark the appropriate option for themselves from the 3 options opposite the question. The first measurement of the scale was as follows; children in the research group: Class 2C answered during the first lesson hour (09:00-09:40). The response time is 40 minutes. Class 3D answered during the second lesson hour (09:50-10:25). The response time is 35 minutes. Class 4D answered during the third lesson hour (10:40-11:10). The response time is 30 minutes. The training was held on March 27, 2024, during the second lesson (09:50-10:30) in a conference hall in the school building with a projector, which was deemed appropriate by the school administration, to facilitate children's participation and to provide a comfortable and quiet environment. The children in the control group took the first measurement of the scale on March 26: 2A class responded during the fourth lesson (11:30-12:10). The response time is 40 minutes. 3A class responded during the fifth lesson (12:50-13:25). The response time is 35 minutes. 4E class responded during the sixth lesson (13:40-14:10). The response time is 30 minutes. The children in the control group (2A, 3A, 4E) took the second measurement of the scale on March 27, 2024, during the first lesson (09:00-09:40) in the conference hall. After the second measurement of the scale was made on March 27, 2024, during the first lesson hour (09:00-09:40), the children in the control group were trained together with the children in the research group in the conference hall during the second lesson hour (09:50-10:30). The second measurement of the scale (2C, 3D, 4D) was administered to the children in the research group on March 27, 27 March 2024 during the third-class hour (10:40-11:20) in the conference hall after the end of the training.

ELIGIBILITY:
Inclusion Criteria:

* The child is 8 to 10 years old,
* The child must be competent to read, understand and answer the items on the scale, and
* It is the parent's consent for their child to participate in the research.

Exclusion Criteria:

* Having a disabled child (mental, hearing, visual, orthopedic, language and speech disability, mental and emotional disease, chronic disease, attention deficit and hyperactivity disorder) and
* The child fills in the scale items incompletely or does not want to fill them in.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Change in hospital perception scale scores of the trained group after training | Immediately after training
  After the planned 40-minute training, the rate of change in children's perception of the hospital was determined with the "Hospital Perception Scale for Healthy Children". An increase in the scale score indicates an increase in the child's negative perception of the hospital.Consisting of 25 items, the total score range of the scale varies between 0 and 50 points. The lowest score that can be obtained from the scale is "0" and the highest score is "50".

CONTACTS AND LOCATIONS:
Overall Officials: Esra ŞAPALOĞLU DÖVENCİ, Principal Investigator — Maltepe University School of Nursing İstanbul, Turkey
Locations (1):
- Esra ŞAPALOĞLU DÖVENCİ, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson ME, Megel ME, Enenbach L, Carlson KL. The voices of children: stories about hospitalization. J Pediatr Health Care. 2010 Mar-Apr;24(2):95-102. doi: 10.1016/j.pedhc.2009.02.008. Epub 2009 Mar 17. PMID 20189061
- [Background] Pelander T, Leino-Kilpi H. Children's best and worst experiences during hospitalisation. Scand J Caring Sci. 2010 Dec;24(4):726-33. doi: 10.1111/j.1471-6712.2010.00770.x. PMID 20487406
- [Background] Canbulat N, Inal S, Sonmezer H. Efficacy of distraction methods on procedural pain and anxiety by applying distraction cards and kaleidoscope in children. Asian Nurs Res (Korean Soc Nurs Sci). 2014 Mar;8(1):23-8. doi: 10.1016/j.anr.2013.12.001. Epub 2013 Dec 14. PMID 25030489
- [Background] Taddio A, Ipp M, Thivakaran S, Jamal A, Parikh C, Smart S, Sovran J, Stephens D, Katz J. Survey of the prevalence of immunization non-compliance due to needle fears in children and adults. Vaccine. 2012 Jul 6;30(32):4807-12. doi: 10.1016/j.vaccine.2012.05.011. Epub 2012 May 19. PMID 22617633
- [Background] Kalmakis KA, Chandler GE. Adverse childhood experiences: towards a clear conceptual meaning. J Adv Nurs. 2014 Jul;70(7):1489-501. doi: 10.1111/jan.12329. Epub 2013 Dec 11. PMID 24329930
- [Background] Li WHC, Chung JOK, Ho KY, Kwok BMC. Play interventions to reduce anxiety and negative emotions in hospitalized children. BMC Pediatr. 2016 Mar 11;16:36. doi: 10.1186/s12887-016-0570-5. PMID 26969158
- [Background] Delvecchio E, Salcuni S, Lis A, Germani A, Di Riso D. Hospitalized Children: Anxiety, Coping Strategies, and Pretend Play. Front Public Health. 2019 Sep 6;7:250. doi: 10.3389/fpubh.2019.00250. eCollection 2019. PMID 31555632
- [Background] Tunc-Tuna P, Acikgoz A. The Effect of Preintervention Preparation on Pain and Anxiety Related to Peripheral Cannulation Procedures in Children. Pain Manag Nurs. 2015 Dec;16(6):846-54. doi: 10.1016/j.pmn.2015.06.006. Epub 2015 Aug 17. PMID 26293196
- [Background] Davidson JE, Aslakson RA, Long AC, Puntillo KA, Kross EK, Hart J, Cox CE, Wunsch H, Wickline MA, Nunnally ME, Netzer G, Kentish-Barnes N, Sprung CL, Hartog CS, Coombs M, Gerritsen RT, Hopkins RO, Franck LS, Skrobik Y, Kon AA, Scruth EA, Harvey MA, Lewis-Newby M, White DB, Swoboda SM, Cooke CR, Levy MM, Azoulay E, Curtis JR. Guidelines for Family-Centered Care in the Neonatal, Pediatric, and Adult ICU. Crit Care Med. 2017 Jan;45(1):103-128. doi: 10.1097/CCM.0000000000002169. PMID 27984278
- [Background] Li HC, Lopez V. Effectiveness and appropriateness of therapeutic play intervention in preparing children for surgery: a randomized controlled trial study. J Spec Pediatr Nurs. 2008 Apr;13(2):63-73. doi: 10.1111/j.1744-6155.2008.00138.x. PMID 18366374
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Tuncay S, Tufekci FG. The effect of nursing interventions with therapeutic play and video animations prepared with psychodrama technique in reducing fear, anxiety, and pain of children at male circumcision: A randomized controlled study. Int J Urol. 2023 Jul;30(7):592-599. doi: 10.1111/iju.15184. Epub 2023 Mar 31. PMID 36999456
- [Background] Ekici B. Development of Hospital Perception Scale for Healthy Children (HPSHC) and Investigation of Its Psychometric Properties. Children (Basel). 2023 Oct 20;10(10):1706. doi: 10.3390/children10101706. PMID 37892369